CLINICAL TRIAL: NCT04807504
Title: A Safety Study of Ropivacaine Concentrations During Continuous Erector Spinae Plane Block for Thoracic Surgery
Brief Title: Ropivacaine Pharmacokinetics in ESP Blocks
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 20G.754
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Local Anesthetic Systemic Toxicity; Pain; Quality of Recovery
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ropivacaine — All patients receive erector spinae plane blocks with ropivacaine.
  Other Names: Naropin

SUMMARY:
This is a pharmacokinetic study to determine risk of local anesthetic systemic toxicity of ropivacaine when used in erector spinae plane blocks for thoracic surgery. Through serial blood sampling and the use of NONMEM population pharmacokinetic analysis this risk will be determined for the study population and other populations as well. Pain and quality of recovery will also be assessed.The erector spinae plane (ESP) block was first described in 2016 as a novel fascial plane block that provided analgesia for thoracic neuropathic pain. Since then hundreds of articles have been published that have reported use of the ESP block for indications such as rib fractures, breast surgery, abdominal surgery, and even shoulder surgery. It has also been studied in thoracic surgery and clinical experience confirms that patients undergoing video-assisted thoracoscopic surgery (VATS) or robot-assisted thoracic surgery experience satisfactory analgesia with ESP blocks. Because the block location is further from the neuraxis than both epidural and paravertebral blocks, ESP blocks have been suggested as a safer alternative to these older blocks but safety data have not yet been generated. In particular, the risk of local anesthetic systemic toxicity (LAST) has not been studied in ESP blocks. While the pharmacokinetics of ropivacaine used for thoracic paravertebral blocks have been established, similar studies have yet to be performed for the newer ESP block. Of particular concern for ESP blocks are two factors not present in some other blocks with established safety: 1). significant intercostal spread has been noted in anatomical studies, which could put patients at risk for LAST and 2). some of the proposed dosing regimens involve the intermittent injection of large bolus doses of local anesthetic. While measurement of arterial plasma levels is useful and necessary to study the safety of ropivacaine given in ESP blocks, the measurements alone do not allow for prediction of plasma levels that would occur in populations as a whole. Nonmem is a population pharmacokinetic application that provides estimates of mean parameters and residual variability in pharmacokinetic values across populations and has been shown to generate better estimates than the two-stage approach. Nonmem will be used in this study to predict pharmacokinetics in populations with different characteristics than the one being studied here, which would create generalizable results.

DETAILED DESCRIPTION:
The erector spinae plane (ESP) block was first described in 2016 as a novel fascial plane block that provided analgesia for thoracic neuropathic pain. Since then hundreds of articles have been published that have reported use of the ESP block for indications such as rib fractures, breast surgery, abdominal surgery, and even shoulder surgery. It has also been studied in thoracic surgery and our clinical experience confirms that patients undergoing video-assisted thoracoscopic surgery (VATS) or robot-assisted thoracic surgery experience satisfactory analgesia with ESP blocks. Because the block location is further from the neuraxis than both epidural and paravertebral blocks, ESP blocks have been suggested as a safer alternative to these older blocks but safety data have not yet been generated. In particular, the risk of local anesthetic systemic toxicity (LAST) has not been studied in ESP blocks. While the pharmacokinetics of ropivacaine used for thoracic paravertebral blocks have been established, similar studies have yet to be performed for the newer ESP block. Of particular concern for ESP blocks are two factors not present in some other blocks with established safety: 1). significant intercostal spread has been noted in anatomical studies, which could put patients at risk for LAST and 2). some of the proposed dosing regimens involve the intermittent injection of large bolus doses of local anesthetic. While measurement of arterial plasma levels is useful and necessary to study the safety of ropivacaine given in ESP blocks, the measurements alone do not allow for prediction of plasma levels that would occur in populations as a whole. Nonmem is a population pharmacokinetic application that provides estimates of mean parameters and residual variability in pharmacokinetic values across populations and has been shown to generate better estimates than the two-stage approach. Nonmem will be used in this study to predict pharmacokinetics in populations with different characteristics than the one being studied here, which would create generalizable results.

ELIGIBILITY:
Inclusion Criteria:

* undergoing robotic or video-assisted thoracic surgery
* able to speak English

Exclusion Criteria:

* active liver disease
* active renal disease
* ropivacaine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with lung cancer, recurrent pneumothoraces, or other condition requiring robotic or video-assisted thoracic surgery are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Mean maximum plasma concentration of ropivacaine | 24 hours

SECONDARY OUTCOMES:
Mean pain scores | 24 hours
  Numerical rating scale pain scores (0-10 where 0 is no pain and 10 is worst pain imaginable)
Opioid consumption | 24 hours
  Mean amount of opioids consumed in morphine milligram equivalents
Sensory levels | 12 hours
  Mean number of dermatomes blocked after erector spinae plane block
Quality of recovery | 24 hours
  The mean quality of recovery 15 survey scores (0-150 where 0 is worst quality of recovery and 150 is best)

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Schwenk, MD, Principal Investigator — Department of Anesthesiology, Sidney Kimmel Medical College at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual data will be shared de-identified upon request

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Karmakar MK, Ho AM, Law BK, Wong AS, Shafer SL, Gin T. Arterial and venous pharmacokinetics of ropivacaine with and without epinephrine after thoracic paravertebral block. Anesthesiology. 2005 Oct;103(4):704-11. doi: 10.1097/00000542-200510000-00008. PMID 16192762
- [Background] Knudsen K, Beckman Suurkula M, Blomberg S, Sjovall J, Edvardsson N. Central nervous and cardiovascular effects of i.v. infusions of ropivacaine, bupivacaine and placebo in volunteers. Br J Anaesth. 1997 May;78(5):507-14. doi: 10.1093/bja/78.5.507. PMID 9175963
- [Background] Luis-Navarro JC, Seda-Guzman M, Luis-Moreno C, Lopez-Romero JL. The erector spinae plane block in 4 cases of video-assisted thoracic surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Apr;65(4):204-208. doi: 10.1016/j.redar.2017.12.004. Epub 2018 Jan 11. English, Spanish. PMID 29336785
- [Derived] Schwenk ES, Lam E, Abulfathi AA, Schmidt S, Gebhart A, Witzeling SD, Mohamod D, Sarna RR, Roy AB, Zhao JL, Kaushal G, Rochani A, Baratta JL, Viscusi ER. Population pharmacokinetic and safety analysis of ropivacaine used for erector spinae plane blocks. Reg Anesth Pain Med. 2023 Sep;48(9):454-461. doi: 10.1136/rapm-2022-104252. Epub 2023 Apr 21. PMID 37085287